CLINICAL TRIAL: NCT02024867
Title: Randomized Non-inferiority Trial of 3 Versus 10 Days of Trimethoprim-Sulfamethoxazole in Community-Associated Skin Abscesses After Surgical Drainage
Brief Title: Evaluation of 3 Versus 10 Days of Antibiotics in Skin Abscesses After Surgical Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucy Holmes, MD (Other)
Collaborators: New York State Department of Health (Other Government); Women & Children's Hospital of Buffalo (Other)
Responsible Party: Sponsor-Investigator, Lucy Holmes, MD, Clinical Associate Professor of Pediatrics, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB 2456
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Skin Disease, Bacterial; Abscess
Keywords: Methicillin resistent Staphylococcus aureus; Staphylococcus aureus
MeSH Terms: conditions — Skin Diseases, Bacterial; Abscess; Staphylococcal Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 days of Trimethoprim-Sulfamethoxazole (Active Comparator): Oral Trimethoprim-Sulfamethoxazole dosed at 10 mg Trimethoprim/kg/day divided twice a day, to a maximum of 640 mg Trimethoprim/day
  Interventions: Drug: Trimethoprim-Sulfamethoxazole
- 3 days of Trimethoprim-Sulfamethoxazole (Experimental): Oral Trimethoprim-Sulfamethoxazole dosed at 10 mg Trimethoprim/kg/day divided twice a day, to a maximum of 640 mg Trimethoprim/day
  Interventions: Drug: Trimethoprim-Sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole — 3 versus 10 days of drug
  Other Names: Septra; Bactrim

SUMMARY:
The objective of this study is to determine if there is a difference in treatment failures and recurrent skin infections when patients are given 3 or 10 days of antibiotics for uncomplicated skin abscesses after they have been surgically drained.

DETAILED DESCRIPTION:
Patients age 3 months to 17 years presenting to a pediatric Emergency Department (ED) with an uncomplicated skin abscess that required surgical drainage were randomized to receive 3 or 10 days of oral trimethoprim-sulfamethoxazole. Patients were evaluated 10 to 14 days later to assess for cure. Patients were contacted 1 month later to determine if they had developed another skin infection. Outcomes were also stratified by methicillin-resistent staphylococcus aureus (MRSA) and methicillin-sensitive staphylococcus aureus (MSSA).

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with a skin abscess that requires surgical drainage (induration ≥ 1 cm in diameter)
* minimally invasive surgical technique with the insertion of a subcutaneous drain can be utilized on the patient

Exclusion Criteria:

* patients requiring immediate hospitalization
* patients who have received 2 or more doses of antibiotics in the previous 36 hours
* patients with diabetes, sickle-cell disease, an immuno-compromising disease, an underlying medical condition predisposing the patient to frequent hospitalizations or medical visits, or indwelling catheters or percutaneous medical devices
* patients with a concurrent, non-abscess infection
* patients with an allergy to Trimethoprim-sulfamethoxazole

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy C Holmes, MD, Principal Investigator — University at Buffalo; Howard Faden, MD, Study Chair — University at Buffalo
Locations (1):
- Women & Children's Hospital of Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Duong M, Markwell S, Peter J, Barenkamp S. Randomized, controlled trial of antibiotics in the management of community-acquired skin abscesses in the pediatric patient. Ann Emerg Med. 2010 May;55(5):401-7. doi: 10.1016/j.annemergmed.2009.03.014. Epub 2009 May 5. PMID 19409657
- [Background] Schmitz GR, Bruner D, Pitotti R, Olderog C, Livengood T, Williams J, Huebner K, Lightfoot J, Ritz B, Bates C, Schmitz M, Mete M, Deye G. Randomized controlled trial of trimethoprim-sulfamethoxazole for uncomplicated skin abscesses in patients at risk for community-associated methicillin-resistant Staphylococcus aureus infection. Ann Emerg Med. 2010 Sep;56(3):283-7. doi: 10.1016/j.annemergmed.2010.03.002. Epub 2010 Mar 26. PMID 20346539
- [Derived] Holmes L, Ma C, Qiao H, Drabik C, Hurley C, Jones D, Judkiewicz S, Faden H. Trimethoprim-Sulfamethoxazole Therapy Reduces Failure and Recurrence in Methicillin-Resistant Staphylococcus aureus Skin Abscesses after Surgical Drainage. J Pediatr. 2016 Feb;169:128-34.e1. doi: 10.1016/j.jpeds.2015.10.044. Epub 2015 Nov 11. PMID 26578074

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 Days; 10 Days: Trimethoprim-Sulfamethoxazole dosed at 10 mg Trimethoprim/kg/day divided twice a day, to a maximum of 640 mg Trimethoprim/day
Period: Overall Study
Arm/Group | 3 Days | 10 Days
Started | 134 | 131
Completed | 125 | 124
Not Completed | 9 | 7
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Days | 10 Days | Total
Number analyzed (Participants) | 125 | 124 | 249
Age, Continuous [Median (Full Range); unit: years] | 4.5 [0.5 to 17] | 3.42 [0.33 to 17] | 4.08 [0.33 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 74 | 157
  Male | 42 | 50 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 17 | 41
  Not Hispanic or Latino | 101 | 107 | 208
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 59 | 122
  White | 49 | 55 | 104
  More than one race | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Abscess location [Number; unit: participants]
  Abscess below the waist | 87 | 91 | 178
  Abscess above the waist | 37 | 30 | 67
  Abscess both locations | 1 | 3 | 4
presence of fever [Number; unit: participants]
  fever | 11 | 11 | 22
  no fever | 114 | 113 | 227
presence of cellulitis [Number; unit: participants]
  cellulitis | 22 | 38 | 60
  no cellulitis | 103 | 86 | 189
Clindamycin administered in ED [Number; unit: participants]
  Yes | 12 | 29 | 41
  No | 113 | 95 | 208
History of abscess [Number; unit: participants]
  Yes | 50 | 42 | 92
  No | 75 | 82 | 157
History of household contact with abscess [Number; unit: participants]
  Yes | 62 | 63 | 125
  No | 63 | 61 | 124
Presence of ≥ 2 Abscesses [Number; unit: participants]
  Yes | 11 | 7 | 18
  No | 114 | 117 | 231
Abscess size [Median (Inter-Quartile Range); unit: cm2] | 6.25 [4 to 12] | 6.25 [4 to 12] | 6.25 [4 to 12]
Culture results [Number; unit: participants]
  MRSA | 69 | 69 | 138
  MSSA | 39 | 40 | 79
  Other | 14 | 14 | 28
  No Growth | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failures
Description: Treatment failures were defined as persistent or increased size of the original abscess requiring further medical or surgical intervention. Treatment cure was defined as no or minimal tenderness, erythema, fever, wound drainage, warmth, fluctuance or induration at the 10 to 14 day follow-up.
Time Frame: up to 2 weeks after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 125 | 124
participants | 9 | 4
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — The sample size of 120 per group was calculated according to an assumed treatment cure rate of 95% with 10 days of antibiotics, and a non-inferiority margin of 7% (allowing up to 88% cure rate with 3 days of antibiotics), to achieve a power of 0.80 (alpha=0.05). An additional 25 patients were recruited to account for an estimated 10% lost to follow-up; p = 0.25, Chi-squared; Rate Difference = 4.0, 95% CI 2-sided [-1.5 to 9.5]

2. Secondary Outcome: Recurrent Skin Infections
Description: Rate of recurrent skin infection among follow-up responders 1 month after enrollment. Patients who were treatment failures were excluded from this analysis since they all received additional medical intervention that could affect the outcome measure.
Time Frame: 1 month after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 115 | 118
participants | 21 | 9
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — described previously; p = 0.02, Chi-squared; Rate Difference = 10.7, 95% CI 2-sided [2.1 to 19.2]

3. Primary Outcome: Treatment Failures Among Patients Infected With Methicillin-Resistant Staphylococcus Aureus
Description: as for outcome 1
Time Frame: up to 2 weeks after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 69 | 69
participants | 8 | 1
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — described previously; p = 0.03, Chi-squared; Rate Difference = 10.1, 95% CI 2-sided [2.1 to 18.2]

4. Primary Outcome: Treatment Failures Among Patients Infected With Methicillin-Sensitive Staphylococcus Aureus
Description: as for outcome 1
Time Frame: up to 2 weeks after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 39 | 40
participants | 1 | 1
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — described previously; p > 0.05, Chi-squared; Rate Difference = 0.1, 95% CI 2-sided [-6.9 to 7.0]

5. Secondary Outcome: Recurrent Skin Infections Among Patients Infected With Methicillin-Resistant Staphylococcus Aureus
Description: as for outcome 2
Time Frame: 1 month after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 60 | 67
participants | 8 | 2
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — described previously; p = 0.046, Chi-squared; Rate Difference = 10.3, 95% CI 2-sided [0.8 to 19.9]

6. Secondary Outcome: Recurrent Skin Infections Among Patients Infected With Methicillin-Sensitive Staphylococcus Aureus
Description: as for outcome 2
Time Frame: 1 month after surgical drainage
Measure: Number; unit: participants
Arm/Group | 3 Days | 10 Days
Number analyzed (Participants) | 38 | 38
participants | 7 | 7
Statistical Analysis 1: Comparison: 3 Days vs 10 Days; Test type: Non-Inferiority or Equivalence — described previously; p > 0.05, Chi-squared; rate difference = 0

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | 3 Days | 10 Days
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/124
Other Adverse Events (participants affected / at risk) | 0/125 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes